CLINICAL TRIAL: NCT03193372
Title: A Study of Patient Concerns and Treatment Satisfaction in Patients Being Treated With Finacea Foam for Rosacea
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19638
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2018-10

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rosacea Concierge Program: Patients diagnosed with rosacea and currently receiving topical monotherapy with Finacea Foam
  Interventions: Drug: Azelaic Acid (Finacea Foam, BAY39-6251)

INTERVENTIONS:
Drug: Azelaic Acid (Finacea Foam, BAY39-6251) — Finacea Foam, Active substance Azelaic acid

SUMMARY:
To survey rosacea patients about their concerns, treatment satisfaction, and quality of life associated with their Finacea Foam treatment

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of rosacea by a medical professional
* Currently using Finacea Foam as topical monotherapy for rosacea
* Willing and able to provide voluntary, informed consent to participate in this study

Exclusion Criteria:

- Use of any other topical treatment for rosacea at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with rosacea and currently receiving topical monotherapy with Finacea Foam
Sampling Method: Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Demographics and clinical characteristics | one-time survey in 2 week recruitment window
  Collected patient demographics and characteristics are :
  * Year of birth
  * Gender
  * Insurance type
Rosacea-relevant comorbidities and complications | one-time survey in 2 week recruitment window
  Patient reported history of the following will be collected :
  * Blepharitis
  * Conjunctivitis
  * Corneal neovascularization/keratitis
  * Depression
  * Migraine
Rosacea subtype | one-time survey in 2 week recruitment window
  Patient reported diagnosis of the following will be collected:
  * Erythematotelangiectatic (facial redness)
  * Papulopustular (bumps and pimples)
  * Phymatous (enlargement of the nose)
  * Ocular (eye irritation)
  * Unknown
Past use of topical rosacea treatments | one-time survey in 2 week recruitment window
  Patient reported use of the following medications will be collected:
  * Metronidazole gel
  * Metronidazole cream
  * Metronidazole lotion
  * Metronidazole emulsion
  * Brimonidine tartrate gel
Patient concerns collected by Rosacea Treatment Preference Questionnaire | one-time survey in 2 week recruitment window
  Rosacea Treatment Preference Questionnaire is a survey to assess patient self-reported rosacea subtype and severity, and to evaluate the concerns that contribute to patient satisfaction/dissatisfaction, as well as treatment decisions with rosacea topical treatments
Treatment satisfaction assessed by Satisfaction with Medicines Questionnaire (SATMED-Q) | one-time survey in 2 week recruitment window
  SATMED-Q is a 17-question, validated, multidimensional generic questionnaire designed for use in patients with any chronic disease treated with medicines
Quality of life measured by Dermatology Life Quality Index (DLQI) | one-time survey in 2 week recruitment window
  DLQI is a widely used dermatology-related quality of life tool

CONTACTS AND LOCATIONS:
Locations (1):
- Xcenda, LLC, Palm Harbor, Florida, United States